CLINICAL TRIAL: NCT04950023
Title: Role of Small Bioactive Molecules in the Progression of Early COPD Diseases
Brief Title: Small Bioactive Molecules in Early COPD Diseases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: LM2021083
Record Dates: First submitted 2021-06-29; First posted 2021-07-02 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-06

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Blood cells and/or pulmonary tissue.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- early COPD: 1) <60 years old; 2) smoking ≥ 10 pack years. 3) with any of the following anomalies: a. Post-bronchodilator FEV1/FVC< 0.7. b. CT image abnormalities: emphysema, air trapping or bronchial wall thickening; c.Rapid decrease of FEV1 (>60 ml/yr).
- Control: 1) <60 years old; 2) Pre-bronchodilator FEV1/FVC≥70% and FEV1 ≥ 80% predicted; 3) no exposure to harmful factors such as cigarettes and dust pollution.

SUMMARY:
To study the predictors contribute to the progression of COPD by follow-up of patients with early COPD and analyze their changes in bioactive molecular, exhaled gas, CT image, lung function, patient's symptoms and life quality.

DETAILED DESCRIPTION:
A research found that nearly 40% of patients with chronic respiratory symptoms who showed significant airway inflammation (airway wall thickening and/or lung structure destruction (emphysema) on chest CT had advanced COPD within 5 years, although their current lung function failed to meet diagnostic criteria for COPD. Current spirometry-based diagnostic methods are not the best predictors of COPD progression and death. CT indicated emphysema and airway inflammation were recognized as better predictors of disease progression and mortality. Based on a large cohort study, some scholars proposed the concept of "early COPD", focusing on people under the age of 50, smoking for more than 10 pack years, having one of the manifestations of early airflow limitation, abnormal chest CT, and rapid decline of FEV1, to study the mechanism of disease progression and early intervention methods.[4] In this study, we enroll participants with early COPD symptoms, to detect the progression of COPD with 3 years of follow-up. The predictors of disease progression and variants of bioactive molecular were analyzed, so as to clarify the progressive mechanism of COPD.

ELIGIBILITY:
Inclusion Criteria:

* 1. <60 years old;

  2. Smoking ≥ 10 pack years.

  3. With any of the following anomalies: a. Post-bronchodilator FEV1/FVC< 0.7. b. CT image abnormalities: emphysema, air trapping or bronchial wall thickening; c.Rapid decrease of FEV1 (>60 ml/yr).

Exclusion Criteria:

* 1. With other known chronic lung diseases, including bronchiectasis, interstitial pulmonary disease, tuberculosis, and pulmonary vascular disease (CTEPH).

  2. With severe pleural disease and/or lesions of the sternum or ribs.

  3. Suffering from serious uncontrolled other systemic diseases, including chest and abdominal surgery, heart attack (angina pectoris, myocardial infarction, malignant arrhythmia, etc.) and cerebrovascular disease (stroke) within 3 months, as well as kidney disease (AKI), cirrhosis, and any malignant tumor except lung cancer.

  4. Suffering from severe cognitive impairment.

  5. With active tuberculosis or are taking anti-tuberculosis treatment.

  6. Pregnancy or lactation.

  7. Previous lung surgery.

  8. Acute upper and lower respiratory system infection within 4 weeks.

Max Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Consecutive eligible patients from Peking University Third Hospital will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2021-05-11 (Actual); Primary Completion 2022-05-11 (Estimated); Study Completion 2024-05-11 (Estimated)

PRIMARY OUTCOMES:
lung function | Lung function will be tested at the 1st year, the 2nd year and the 3rd year.
  Patients' lung function will be tested to identify air flow decrease in the early COPD group and the control group.

SECONDARY OUTCOMES:
Blood samples | The 1st year and the 3rd year of follow-up
  Collect venous blood to detect cytokines and other molecular.
CT | The 1st year and the 3rd year of follow-up
  Both inspiration phase and expiration phase are required
Exhaled breath condensate | The 1st year and the 3rd year
  Using commercially available exhaled breath condensate collection
Exhaled hydrogen sulfide and nitric oxide | The 1st year and the 3rd year
  Using breath analyzer to detect real-time release
Pulmonary tissue | The 1st year patients are enrolled
  Pulmonary tissue will be obtained from patients who are about to undergo resection, for example, COPD patients with lung cancer.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martinez FJ, Han MK, Allinson JP, Barr RG, Boucher RC, Calverley PMA, Celli BR, Christenson SA, Crystal RG, Fageras M, Freeman CM, Groenke L, Hoffman EA, Kesimer M, Kostikas K, Paine R 3rd, Rafii S, Rennard SI, Segal LN, Shaykhiev R, Stevenson C, Tal-Singer R, Vestbo J, Woodruff PG, Curtis JL, Wedzicha JA. At the Root: Defining and Halting Progression of Early Chronic Obstructive Pulmonary Disease. Am J Respir Crit Care Med. 2018 Jun 15;197(12):1540-1551. doi: 10.1164/rccm.201710-2028PP. No abstract available. PMID 29406779